CLINICAL TRIAL: NCT03104894
Title: The Effect of Meibomian Glands Massage on Signs and Symptoms of Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barzilai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0137-13-BRZ
Record Dates: First submitted 2017-03-14; First posted 2017-04-07 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-04

CONDITIONS: MGD-Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: patient will be assigned to the study/control group by randomization soft ware. The results will be documented and kept by the doctor who preforms the meibomian glands massage/ sham massage. All patients will receive study number. Follow up examination will be preformed by another doctor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): The study group will receive meibomian glands massage and artificial drops PRN
  Interventions: Procedure: Meibomian Glands Massage; Device: Meibomian Massage device
- Control Group (Sham Comparator): The control group will receive sham meibomian glands massage and artificial drops PRN.
  Interventions: Procedure: Sham Meibomian Glands Massage

INTERVENTIONS:
Procedure: Meibomian Glands Massage — Meibomian gland expression
  Arms: Study Group
Procedure: Sham Meibomian Glands Massage — Touching the eyelids gently
  Arms: Control Group
Device: Meibomian Massage device — Meibomian glands expression with applicator
  Arms: Study Group

SUMMARY:
The study aims to investigate whether combined treatment of MGD massage and artificial tears will improve signs and symptoms of dry eye compared to artificial tears alone.

The meibomian glands secrete meibum which is the oily component of the tear film layer. The meibum plays a pivotal role in preventing tear evaporation and smoothening the tears film .

Meibomian gland dysfunction is a common condition that affects 39%-50% of the population. It is part of inflammatory disease of the eyelids called blepharitis. Associated syndromes are rosacea and dry eye syndrome .

Sign and symptoms are: irritation, hyperemia, burning sensation, photophobia, epiphora and blur.

Spectrometry analysis shows change it the fatty acids conformation such as increase in levels of branched-chain fatty acids and decrease in saturated fatty acids .

Subsequently the clotted meibum results in glands blockage that can be graded in 0-4 grade scale: grade 2- meibum secretion thick and oily, grade 3- meibum secretion granular-toothpaste like.

Although MGD is not often accompanied with inflammatory signs it is a common cause for evaporative dry eye.

DETAILED DESCRIPTION:
In order to investigate the relation between meibomian gland massage outcomes and signs and symptoms of dry eye, randomized prospective study will be conducted. Patients, who arrive to Barzilai Medical Center out patients' clinic, are diagnosed with MGD 2-3 and signed informed consent form shall be included in the trial, then randomized to study group or control group.

The study group will receive meibomian glands massage and artificial drops PRN, whereas the control group will receive sham massage and artificial drops. Each visit at the clinic will include dry examinations and questionnaire.

Follow up examination are due after one week, monthly visits up to 4 months, then after half year, 8 months and one year.

Statistical methods: in order to evaluate to treatment effect T-Test analysis will be calculated, significant result is when P<0.05.

Data will be recorded into to electronic sheets. Subjects' confidentiality will be assured by masking any identifying details and a random number will be assigned prior results analysis stage

ELIGIBILITY:
Inclusion Criteria:

* Adult Individuals (age≥18Y) with MGD levels 2-3 that are capable to make an informed decision about their participation in the trial.

Exclusion Criteria:

* pregnant women, subjects who received prior Meibomian gland massage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-08; Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Improvement in Tear Break up Time TBUT. | 1 month
  Tear break up time will be measured in seconds. The score is expected to be higher.
Improvement in Ocular Surface Disease Index questionnaire score (OSDI) | 1 month
  OSDI score will be calculated according a formula: (sum of scores) X 25 divided by the number of questions answered. The score is expected to be lower.

CONTACTS AND LOCATIONS:
Locations (1):
- Barzilai Medical Center, Ashkelon, Is, Israel

IPD SHARING:
Plan to Share IPD: No